CLINICAL TRIAL: NCT04289077
Title: The Evaluation of Health-related Quality of Life Issues Experienced by Patients With Desmoid-type Fibromatosis
Brief Title: Quality of Life of Patients With Desmoid-type Fibromatosis
Acronym: QUALIFIED
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: Radboud University Medical Center (Other); The Netherlands Cancer Institute (Other); Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, C. Verhoef, Prof. dr. C. Verhoef, MD, PhD, Erasmus Medical Center
Other Study IDs: MEC-2019-0816
Record Dates: First submitted 2020-02-24; First posted 2020-02-28 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Desmoid Tumor; Desmoid-type Fibromatosis
Keywords: Health-related quality of life; Quality of life
MeSH Terms: conditions — Desmoid Tumors | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with histopathological proven DTF
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — - Baseline questionnaire, version 1.0, October 29 2019, (Dutch) - Health care utilization, version 1.0, October 29 2019, (Dutch) - Decision-making, version 1.0, October 29 2019, (Dutch) - EORTC QLQ-C30, version 3.0, (Dutch) - DTF-QoL, version 1.0, October

SUMMARY:
Rationale: Desmoid-type fibromatosis (DTF) is a rare, histologically benign, soft tissue tumour. Although incapable of metastasizing, the clinical course is unpredictable and can be aggressive because of local invasive growth. Various treatments are available including; surgical resection, radiotherapy, hormonal therapy and chemotherapy. Nowadays there is a trend towards a more conservative strategy with a wait and see policy because of high recurrence rates after surgical resection. Health-related quality of life (HRQL) is a corner stone in treatment choice and can be used during the disease for monitoring the impact of the disease on physical, psychological and social level. Additionally, HRQL can be in important endpoint for future clinical trials. Today, no HRQL-tools are available which capture the needs of DTF patients. The hypothesis is that patients with DTF have issues on several HRQL domains including physical, social and emotional well-being. For this reason we developed a list of items based on previous research. This study aims to evaluate HRQL issues experienced by DTF patients.

Purpose: Multi-centre, cross-sectional, observational study to measure HRQL of DTF patients and to evaluate the prevalence of the experienced problems.

DETAILED DESCRIPTION:
Objectives: The primary objective is to evaluate HRQoL problems in adult DTF patients. The secondary objectives are: 1) to compare the level of HRQoL of DTF patients to the general population, 2) to identify patient subgroups who are at risk for developing certain HRQoL problems, 3) to evaluate patient preferences regarding their health care needs for DTF.

Outline: All patients, aged above 18 years, with a histopathological proved DTF tumour and sufficient Dutch language skills who have received their last check-up in the hospital within the last five years (April 2014). Patients treated in one of the participating centres, will be asked to fill out a set of questionnaires (baseline questionnaire, health care utilization, decision making, EORTC QLQ-C30, DTF-specific questionnaire, and the EQ-5D-5L). Patients will only have to fill out these questionnaires once.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older
* Histopathological proven DTF, regardless of disease stage or treatment.
* Diagnosed between January 1990 and July 2020, with a visit to the hospital for their DTF (between October 2014 and July 2020)
* Sufficient Dutch language skills
* Competent to complete a questionnaire
* Written informed consent

Exclusion Criteria:

• Familial adenomatous polyposis (FAP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients, aged ≥18 years, diagnosed with a histopathological proven DTF, regardless of disease stage and received treatment(s) who have received their last check-up of their DTF in one of the participating hospitals the hospital between October 2014 and July 2020.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2020-08-06 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
EORTC QLQ-C30 questionnaire (European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire-Core-30; version 3.0) | Participants have to fill out the questionnaire once and have to complete the questionnaire within 3 months after the invitation. A reminder for participation will be send one month after the initial invitation.
  Each question will be scored: not at all (1), a little (2), quite a bit (3), very much (4). The scores of the EORTC-QLQ30 will be calculated using a Likert scale from 1-4. The scoring manual of the EORTC will be followed. After linear transformation, all scales and single item measures range in score from 0-100. Scores for each scale will be reported as mean (SD), or as median (IQR). A higher score on the functional scales and global quality of life means better functioning and HRQoL, whereas a higher score on the symptom scales means more complaints. The EORTC QLQ-C30 summary score will be calculated using the mean scores of the function scales and the reversed mean scores of the symptom scales and represented as the mean of the combined 13 QLQ-C30 scale scores (financial impact and global health status excluded). A higher summary score represented a better outcome.
DTF-QoL questionnaire (Desmoid-type fibromatosis Quality of Life Questionnaire) | Participants have to fill out the questionnaire once and have to complete the questionnaire within 3 months after the invitation. A reminder for participation will be send one month after the initial invitation.
  The scores for each item of the DTF-QoL will be calculated using a Likert scale from 1-4. The scores of each item will be calculated as mean ± SD, or as median (IQR). These scores (median or mean) will be reported per item.
EQ-5D-5L questionnaire (EuroQol five-dimensional questionnaire; version 1.0) | Participants have to fill out the questionnaire once and have to complete the questionnaire within 3 months after the invitation. A reminder for participation will be send one month after the initial invitation.
  Measures health-related quality of life on five dimensions of health: mobility, self-care, usual activities, pain-discomfort, and anxiety/depression. Additionally two questions aim to rank a patients' health (scale 0-100, with 100 representing a better health). Each of the five dimensions can be divided into five levels of perceived problems: no problems (level 1), slight problems (level 2), moderate problems (level 3), severe problems (level 4) and extreme problems (level). Health states can be converted into single index values. The outcomes will be reported as frequency (proportion) of reported problems for each level and for each dimension. The Visual Analogue Scale (VAS) data will be presented as a mean value (SD). In case of skewed data, median values and IQR will be used.

SECONDARY OUTCOMES:
EORTC QLQ-C30 questionnaire (European Organisation for Research and Treatment of Cancer, Quality of Life Questionnaire-Core-30; version 3.0) | Participants have to fill out the questionnaire once and have to complete the questionnaire within 3 months after the invitation. A reminder for participation will be send one month after the initial invitation.
  See primary outcome 1 for a detailed description of the EORTC QLQ-C30 questionnaire.
  The median or mean values for each scale of the EORTC QLQ-C30 from DTF patients will be compared to the median or mean scores per scale of the general population.
Baseline questionnaire (version 1.0) | Participants have to fill out the questionnaire once and have to complete the questionnaire within 3 months after the invitation. A reminder for participation will be send one month after the initial invitation.
  Subgroups will be created based on the information of the baseline questionnaire and will encompass: sex (male, female), age groups (categorized based by the median age and/or quartiles), primary treatment type (surgical resection, systemic treatment, radiotherapy, local treatment (e.g. cryoablation), ethnicity, educational level, relationship status, job demands, comorbidities, tumour location, and tumour recurrences.
  Outcomes of this questionnaire will be descriptive and are expressed as numbers with corresponding percentages.
  Mean or median scores of each scale (EORTC QLQ-C30, version 3.0), items (DTF-QoL, version 1,0) or frequency scores (EQ-5D-5L, version 1,0) will be calculated for each relevant subgroup.
Healt care utilization questionnaire (version 1.0) | Participants have to fill out the questionnaire once and have to complete the questionnaire within 3 months after the invitation. A reminder for participation will be send one month after the initial invitation.
  The health care utilization questionnaire contains the following topics: satisfaction with received care, frequency of visits to the general practitioner / specialist, satisfaction with the follow-up schedule, preferences and needs for receiving care in a DTF expert centre, receiving additional care of support from professionals (medical and non-medical). Outcomes will be descriptive and reported in numbers and corresponding frequencies per answer option.
Decision making questionnaire (version 1.0) | Participants have to fill out the questionnaire once and have to complete the questionnaire within 3 months after the invitation. A reminder for participation will be send one month after the initial invitation.
  Six questions were designed to obtain information on how patients make medical decisions, what their current role is and what their preferred role, and one question regarding their awareness of their choices, the benefits and risks of certain treatment and whether they received support an advice are designed. Two questions were designed to gain insight into the reasons for choosing an active form of treatment.
  Outcomes of this questionnaire will be descriptive and expressed as numbers with corresponding percentages.

CONTACTS AND LOCATIONS:
Overall Officials: C. Verhoef, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (4):
- Netherlands (3):
  - 3. Antoni van Leeuwenhoek Ziekenhuis (AVL) / The Netherlands Cancer Instituut , Amsterdam, The Netherlands, Amsterdam
  - Radboud University Medical Center (MC), Nijmegen, The Netherlands, Nijmegen
  - Erasmus MC Cancer Institute, Rotterdam
- Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kasper B, Baumgarten C, Garcia J, Bonvalot S, Haas R, Haller F, Hohenberger P, Penel N, Messiou C, van der Graaf WT, Gronchi A; Desmoid Working Group. An update on the management of sporadic desmoid-type fibromatosis: a European Consensus Initiative between Sarcoma PAtients EuroNet (SPAEN) and European Organization for Research and Treatment of Cancer (EORTC)/Soft Tissue and Bone Sarcoma Group (STBSG). Ann Oncol. 2017 Oct 1;28(10):2399-2408. doi: 10.1093/annonc/mdx323. PMID 28961825
- [Background] Posner MC, Shiu MH, Newsome JL, Hajdu SI, Gaynor JJ, Brennan MF. The desmoid tumor. Not a benign disease. Arch Surg. 1989 Feb;124(2):191-6. doi: 10.1001/archsurg.1989.01410020061010. PMID 2916941
- [Background] Crago AM, Denton B, Salas S, Dufresne A, Mezhir JJ, Hameed M, Gonen M, Singer S, Brennan MF. A prognostic nomogram for prediction of recurrence in desmoid fibromatosis. Ann Surg. 2013 Aug;258(2):347-53. doi: 10.1097/SLA.0b013e31828c8a30. PMID 23532110
- [Background] Gronchi A, Colombo C, Le Pechoux C, Dei Tos AP, Le Cesne A, Marrari A, Penel N, Grignani G, Blay JY, Casali PG, Stoeckle E, Gherlinzoni F, Meeus P, Mussi C, Gouin F, Duffaud F, Fiore M, Bonvalot S; ISG and FSG. Sporadic desmoid-type fibromatosis: a stepwise approach to a non-metastasising neoplasm--a position paper from the Italian and the French Sarcoma Group. Ann Oncol. 2014 Mar;25(3):578-583. doi: 10.1093/annonc/mdt485. Epub 2013 Dec 9. PMID 24325833
- [Background] Gundle KR, Cizik AM, Jones RL, Davidson DJ. Quality of life measures in soft tissue sarcoma. Expert Rev Anticancer Ther. 2015 Jan;15(1):95-100. doi: 10.1586/14737140.2015.972947. Epub 2014 Nov 7. PMID 25377073
- [Background] Gounder MM, Mahoney MR, Van Tine BA, Ravi V, Attia S, Deshpande HA, Gupta AA, Milhem MM, Conry RM, Movva S, Pishvaian MJ, Riedel RF, Sabagh T, Tap WD, Horvat N, Basch E, Schwartz LH, Maki RG, Agaram NP, Lefkowitz RA, Mazaheri Y, Yamashita R, Wright JJ, Dueck AC, Schwartz GK. Sorafenib for Advanced and Refractory Desmoid Tumors. N Engl J Med. 2018 Dec 20;379(25):2417-2428. doi: 10.1056/NEJMoa1805052. PMID 30575484
- [Background] Husson O, Younger E, Dunlop A, Dean L, Strauss DC, Benson C, Hayes AJ, Miah A, van Houdt W, Zaidi S, Smith M, Williams J, Jones RL, van der Graaf WTA. Desmoid fibromatosis through the patients' eyes: time to change the focus and organisation of care? Support Care Cancer. 2019 Mar;27(3):965-980. doi: 10.1007/s00520-018-4386-8. Epub 2018 Aug 28. PMID 30155568
- [Background] van Broekhoven DL, Grunhagen DJ, den Bakker MA, van Dalen T, Verhoef C. Time trends in the incidence and treatment of extra-abdominal and abdominal aggressive fibromatosis: a population-based study. Ann Surg Oncol. 2015 Sep;22(9):2817-23. doi: 10.1245/s10434-015-4632-y. Epub 2015 Jun 5. PMID 26045393
- [Background] Bonvalot S, Ternes N, Fiore M, Bitsakou G, Colombo C, Honore C, Marrari A, Le Cesne A, Perrone F, Dunant A, Gronchi A. Spontaneous regression of primary abdominal wall desmoid tumors: more common than previously thought. Ann Surg Oncol. 2013 Dec;20(13):4096-102. doi: 10.1245/s10434-013-3197-x. Epub 2013 Sep 20. PMID 24052312
- [Background] Penel N, Le Cesne A, Bonvalot S, Giraud A, Bompas E, Rios M, Salas S, Isambert N, Boudou-Rouquette P, Honore C, Italiano A, Ray-Coquard I, Piperno-Neumann S, Gouin F, Bertucci F, Ryckewaert T, Kurtz JE, Ducimetiere F, Coindre JM, Blay JY. Surgical versus non-surgical approach in primary desmoid-type fibromatosis patients: A nationwide prospective cohort from the French Sarcoma Group. Eur J Cancer. 2017 Sep;83:125-131. doi: 10.1016/j.ejca.2017.06.017. Epub 2017 Jul 20. PMID 28735069
- [Background] Timbergen MJM, van de Poll-Franse LV, Grunhagen DJ, van der Graaf WT, Sleijfer S, Verhoef C, Husson O. Identification and assessment of health-related quality of life issues in patients with sporadic desmoid-type fibromatosis: a literature review and focus group study. Qual Life Res. 2018 Dec;27(12):3097-3111. doi: 10.1007/s11136-018-1931-3. Epub 2018 Jul 16. PMID 30014458
- [Background] Nolte S, Liegl G, Petersen MA, Aaronson NK, Costantini A, Fayers PM, Groenvold M, Holzner B, Johnson CD, Kemmler G, Tomaszewski KA, Waldmann A, Young TE, Rose M; EORTC Quality of Life Group. General population normative data for the EORTC QLQ-C30 health-related quality of life questionnaire based on 15,386 persons across 13 European countries, Canada and the Unites States. Eur J Cancer. 2019 Jan;107:153-163. doi: 10.1016/j.ejca.2018.11.024. Epub 2018 Dec 19. PMID 30576971
- [Background] Giesinger JM, Kieffer JM, Fayers PM, Groenvold M, Petersen MA, Scott NW, Sprangers MA, Velikova G, Aaronson NK; EORTC Quality of Life Group. Replication and validation of higher order models demonstrated that a summary score for the EORTC QLQ-C30 is robust. J Clin Epidemiol. 2016 Jan;69:79-88. doi: 10.1016/j.jclinepi.2015.08.007. Epub 2015 Sep 28. PMID 26327487
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet. 2007 Oct 20;370(9596):1453-7. doi: 10.1016/S0140-6736(07)61602-X. PMID 18064739

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-26): https://cdn.clinicaltrials.gov/large-docs/77/NCT04289077/Prot_SAP_000.pdf